CLINICAL TRIAL: NCT06403527
Title: Ultrasound Guyded Venous Puncture for Safe AF Ablation Procedures
Acronym: ULYSSES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB recommendation
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ULYSSES
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Puncture for Safe Atrial Fibrillation Ablation
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, prospective, randomized, interventional, multicenter trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Active Comparator): Ultrasound guided venous access during AF ablation
  Interventions: Other: Ultrasound guided venous access during AF ablation
- Control (No Intervention): Conventional venous puncture guided by palpation

INTERVENTIONS:
Other: Ultrasound guided venous access during AF ablation — Ultrasound guided venous access during AF ablation
  Other Names: Ultrasound
  Arms: Interventional arm

SUMMARY:
To assess if ultrasound guided venous puncture reduces the risk for access site complication in the contex of atrial fibrillation ablation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Age ≥18 years
  2. Signed written informed consent
  3. Planned transvenous catheter ablation procedure for AF or left atrial tachycardia
  4. Willingness to participate in follow-up

Exclusion Criteria

1. Patient is unable or unwilling to provide informed consent
2. Planned/required arterial access (e.g. for blood pressure monitoring)
3. Patient has contra-indication to oral anticoagulation
4. Known coagulation disorder or Thrombocytopenia <150.000/ul.

6. Women currently pregnant or breastfeeding or women of childbearing potential without highly effective contraception (PEARL-Index < 1%), 7. Patient is included in another clinical trial 8. Inability to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1075 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2026-02-04 (Actual); Study Completion 2026-02-04 (Actual)

PRIMARY OUTCOMES:
occurrence of venous access site complications | 30 days
  occurrence of venous access site complications until 30 days after the procedure defined as AV fistula, false aneurysm or access site bleeding requiring intervention (BARC 3 A or higher)

CONTACTS AND LOCATIONS:
Overall Officials: Neda Tarighi, Doctor, Study Chair — CCB
Locations (1):
- Boris Schmidt, Frankfurt am Main, Hesse, Germany